CLINICAL TRIAL: NCT01059474
Title: Transdermal Absorption of DMPS and Its Effect on Urinary Mercury Excretion
Brief Title: Transdermal Absorption of Dimercaptopropane-1-Sulfonate (DMPS) and Effect on Urinary Mercury Excretion
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Banner Health (Other)
Collaborators: Phoenix Children's Hospital (Other)
Responsible Party: Anne-Michelle Ruha, M.D., Banner Health
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DMPS 09-125
Record Dates: First submitted 2010-01-19; First posted 2010-02-01 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-05

CONDITIONS: Toxicity
Keywords: DMPS; mercury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DMPS (Experimental): We will recruit 10 healthy adult volunteers, over 18 years of age, who eat at least three servings of fish per week (since this diet is associated with detectable levels of mercury in the urine which may rise following chelation). Patients with known allergies to DMPS or sulfa drugs or history of neurologic or renal disease will be excluded. We will also control for number of mercury containing dental amalgams. History will be obtained regarding any potential mercury exposures or recent vaccinations.
  Interventions: Drug: transdermal DMPS

INTERVENTIONS:
Drug: transdermal DMPS — 12 hr urine mercury and creatinine levels will be measured on all volunteers prior to any treatment. The urine will be collected in acid-washed or heavy-metal-free specialty containers. Each volunteer will then receive 120 mg of transdermal DMPS, applied to the bicep area of one arm. The area of application will not exceed 2% body surface area. After dosing, urine will be collected for the next 12 hours (using the same protocol and send-out procedure) and assayed for mercury and creatinine levels.
  Additionally, after dosing, an intravenous catheter will be placed in the arm of each subject for blood draws. Blood samples will be obtained at 30 minutes, 60 minutes, 90 minutes, 2 hours, 4 hours and 6 hours after application of the DMPS.

SUMMARY:
DMPS is a metal chelator which is approved for use in Europe. While not an FDA-approved drug in the US, it is easily obtained and administered by alternative health practitioners to their patients. A formulation called 'TD DMPS' (transdermal DMPS) is in use, despite the fact there is no published literature to support that the agent is absorbed transdermally. The investigators hypothesis is that DMPS is not absorbed through the skin. The investigators plan to apply TD DMPS to healthy volunteers and then test serum for presence of DMPS. In addition the investigators will measure urinary mercury concentrations pre and post DMPS application.

DETAILED DESCRIPTION:
I. Background Information and Literature:

2,3-dimercaptopropane-1-sulfonate (DMPS) is a chelating agent that has been used for years in Europe for treatment of poisoning by metals such as mercury, arsenic, and lead. It is a water soluble analog of dimercaptopropanol (British anti-Lewisite, or BAL), which is an FDA approved chelating agent administered via deep intramuscular injection. DMPS is not FDA approved, but is approved in Europe and is available in Germany without a prescription, as Dimaval. It is felt to have less toxicity than BAL, and unlike BAL, is effective when administered orally(1).

A comprehensive review by Aposhian, et al (1) notes that DMPS has been studied since the late 1950's in the Soviet Union and China and appears innocuous. This review mentions a 1979 study which followed 168 scleroderma patients receiving DMPS for 10 years. Some patients experienced mild side effects such as minor allergic reaction (26 patients, none with anaphylaxis), nausea (11 patients), vertigo (7 patients), weakness (4 patients), or itching (3 patients). No renal toxicity was noted. Additionally, chelation therapy with oral DMPS was found to be safe when used in a series of patients with methylmercury toxicity from contaminated grain in Iraq in 1972 (2). It was also not associated with any adverse effects when used to orally chelate lead poisoned children in Baltimore, Maryland in 1985 (3). This 1985 study cites case series of DMPS being safely and effectively used for treatment of lead poisoning and inorganic mercury poisoning as well.

DMPS showed no mutagenicity in the Ames salmonella microsome plate test.

Soviet studies showed that when their usual human dose of 5mg/kg IV was increased to 100mg/kg IV, ulceration or necrosis at the injection site was noted. Animal studies with very large (50mg/kg) IV doses showed tremors, tachycardia, dyspnea, vomiting, and defecation. Other animal studies, however, noted no behavioral, weight, or blood composition changes in animals given 15 or 80mg/kg IV DMPS.

Animal and human data demonstrated DMPS to be less toxic than the currently FDA approved chelating agent, BAL (1).

Our study proposes to apply a single dose of a liquid formulation of DMPS to the skin. Though there is no available animal or human data on this form of application, it is being used throughout the U.S. by many naturopaths and physicians as a chelating agent for children with autism. In the pamphlets and protocols of these physicians, the only side effects they mention seeing are mild skin rash and, with chronic therapy, possible depletion of other necessary metals (such as zinc and magnesium), for which they provide a mineral supplement.

Since we will be using a small, one-time only dose, there is no risk of significant metal or mineral depletion. The main risk to subjects will be mild skin rash, which can easily be monitored.

II. Manufacturing information:

The transdermal DMPS to be used in the study will be obtained from Bellevue Pharmacy, a compounding pharmacy (1034 S. Brentwood Blvd. Suite 102 St. Louis, MO 63117), which supplies this product to doctors all over the U.S. According to the literature they provide, the product is an anhydrous gel dispensed in 30 ml bottles. Each drop reportedly contains 1mg of DMPS and 4mg of glutathione. We will buy the product we need for the study in one bulk batch since each subject will only be getting one dose.

Prior to conducting the study, a bottle will be sent to the FDA lab to be analyzed for confirmation of the presence of DMPS in the gel.

III. Investigator Qualifications:

Principal Investigator:

Anne-Michelle Ruha, MD, FACMT

Assistant Investigator:

Jennifer Smith, MD

Both investigators are board certified emergency physicians, Dr. Ruha is a board certified medical toxicologist, and Dr. Smith is near completion of her fellowship in medical toxicology (see attached curriculum vitae). At least one investigator will be present at all times during the application of the product and the follow-up blood draws. We will be prepared to deal with any acute reactions which occur, allergic or otherwise. After this time period we will be available by phone via the poison center 24 hours a day, 7 days a week for any concerns or complications experienced by study subjects.

IV. Study Protocol:

Since transdermal DMPS delivery is widely used but has not been studied, the clinical question we wish to answer is whether DMPS is absorbed through the skin after transdermal application and if so, whether it increases urinary mercury excretion.

We will recruit 10 healthy adult volunteers, over 18 years of age, who eat at least three servings of fish per week (since this diet is associated with detectable levels of mercury in the urine which may rise following chelation). Patients with known allergies to DMPS or sulfa drugs or history of neurologic or renal disease will be excluded. We will also control for number of mercury containing dental amalgams. History will be obtained regarding any potential mercury exposures or recent vaccinations.

12 hr urine mercury and creatinine levels will be measured on all volunteers prior to any treatment. The urine will be collected in acid-washed or heavy-metal-free specialty containers. It will be refrigerated during and after the collection period and shipped to NMS labs (with cooling pack) for measurement of mercury levels and mercury:creatinine ratios. Each volunteer will then receive 120 mg of transdermal DMPS, applied to the bicep area of one arm. The area of application will not exceed 2% body surface area. The dose of DMPS was determined based on the "challenge dose" from the "Buttar Autism treatment Protocol", used by Dr. Rashid Buttar in his clinic for the treatment of autistic children. This protocol advises use of 3 mg/kg, with a max dose of 120 mg. After dosing, urine will be collected for the next 12 hours (using the same protocol and send-out procedure) and assayed for mercury and creatinine levels.

Additionally, after dosing, an intravenous catheter will be placed in the arm of each subject for blood draws. Blood samples will be obtained at 30 minutes, 60 minutes, 90 minutes, 2 hours, 4 hours and 6 hours after application of the DMPS. These samples will be sent to the FDA for DMPS analysis.

Subjects will be monitored during application and for the subsequent 6 hours for the development of skin rash or any other symptoms related to the DMPS, though this is unlikely. If rash develops the skin will be washed and the reaction can be treated as necessary. At the end of the 6 hours, the skin will be cleansed with soap and water and the treatment period ends.

When analyzing the data after collection, we will first look at whether any DMPS was detectable in the blood after application. If so, we will examine the 12 hour urine mercury levels from before and after application to determine whether this increased. We will control for number of dental amalgams, which can affect baseline urinary Hg levels. If an increase is detected, we will compare the magnitude of this increase to available data on urinary Hg excretion increase after oral DMPS administration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult

Exclusion Criteria:

* Under 18 years of age
* Allergy to sulfa
* Eat less than three fish servings per week

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2010-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
serum DMPS level | within 6 hours of application

SECONDARY OUTCOMES:
change in urinary mercury excretion | 12 hours preceeding and following DMPS

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Michelle Ruha, M.D., Principal Investigator — Banner Health
Locations (1):
- Department of Medical Toxicology, Phoenix, Arizona, United States

REFERENCES:
- [Background] Aposhian HV. DMSA and DMPS--water soluble antidotes for heavy metal poisoning. Annu Rev Pharmacol Toxicol. 1983;23:193-215. doi: 10.1146/annurev.pa.23.040183.001205. No abstract available. PMID 6307120
- [Background] Clarkson TW, Magos L, Cox C, Greenwood MR, Amin-Zaki L, Majeed MA, Al-Damluji SF. Tests of efficacy of antidotes for removal of methylmercury in human poisoning during the Iraq outbreak. J Pharmacol Exp Ther. 1981 Jul;218(1):74-83. PMID 7241391
- [Background] Chisolm JJ Jr, Thomas DJ. Use of 2,3-dimercaptopropane-1-sulfonate in treatment of lead poisoning in children. J Pharmacol Exp Ther. 1985 Dec;235(3):665-9. PMID 4078728
- [Background] Aposhian HV. Mobilization of mercury and arsenic in humans by sodium 2,3-dimercapto-1-propane sulfonate (DMPS). Environ Health Perspect. 1998 Aug;106 Suppl 4(Suppl 4):1017-25. doi: 10.1289/ehp.98106s41017. PMID 9703487
- [Background] Gross L. A broken trust: lessons from the vaccine--autism wars. PLoS Biol. 2009 May 26;7(5):e1000114. doi: 10.1371/journal.pbio.1000114. Epub 2009 May 26. PMID 19478850
- [Background] Torres-Alanis O, Garza-Ocanas L, Bernal MA, Pineyro-Lopez A. Urinary excretion of trace elements in humans after sodium 2,3-dimercaptopropane-1-sulfonate challenge test. J Toxicol Clin Toxicol. 2000;38(7):697-700. doi: 10.1081/clt-100102382. PMID 11192456